CLINICAL TRIAL: NCT07376473
Title: Psychometric Validation of the MQOL-FR and Descriptive Assessment of Quality of Life in Patients With Meningiomas
Acronym: MenQOL 2
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Other Study IDs: D25-P039
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Intracranial Meningioma; Meningioma; Health-related Quality of Life
Keywords: meningioma; intracranial meningioma; quality of life; health-related quality of life; HRQoL; patient-reported outcomes; PRO; questionnaire validation; psychometric validation; MQOL; FACT-Br; EQ-5D-5L; REDCap; neurosurgery
MeSH Terms: conditions — Meningioma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Meningioma cohort: Adults (≥18 years) with intracranial meningioma diagnosed on imaging and/or confirmed surgically. Participants complete a single online, self-administered questionnaire session via a secure REDCap link. There is no study-related treatment, no additional visit, and usual care is unchanged.
  Interventions: Other: Quality-of-life questionnaire administration

INTERVENTIONS:
Other: Quality-of-life questionnaire administration — Single-session completion of patient-reported outcome questionnaires: MQOL-FR (meningioma-specific), EQ-5D-5L, and FACT-Br, administered online via REDCap (approximately 30-45 minutes; may be completed in multiple sittings).

SUMMARY:
This non-interventional study aims to validate the French version of a meningioma-specific quality-of-life questionnaire (MQOL-FR) and to describe health-related quality of life in adults diagnosed with an intracranial meningioma.

Participants will be invited to complete online questionnaires through a secure REDCap link. After reading the study information and recording their non-opposition, participants will complete: (1) MQOL-FR (meningioma-specific), (2) EQ-5D-5L (generic health-related quality of life), and (3) FACT-Br (brain tumor-specific quality of life). The questionnaire session takes approximately 30-45 minutes and can be completed in more than one sitting using a REDCap access code. There is no additional visit and no change in usual care.

The study will recruit adults (≥18 years) with a meningioma diagnosis based on imaging and/or confirmed by surgery, through the GHU Paris-Sainte-Anne neurosurgery clinic and through patient/community networks. The goal is to obtain 100 fully completed MQOL-FR questionnaires suitable for psychometric analyses.

DETAILED DESCRIPTION:
Meningiomas are common intracranial tumors and may substantially affect psychological, social, and functional well-being, including in patients managed conservatively. However, validated meningioma-specific quality-of-life tools are limited. The MQOL questionnaire was originally developed as a patient-centered, meningioma-specific instrument; a prior French translation/adaptation and pilot evaluation has been conducted. This study (MenQOL2) is designed to complete an in-depth psychometric validation of the French version (MQOL-FR) in a larger cohort and to provide a descriptive assessment of quality of life in French patients with meningioma.

This is a single-center, non-interventional, questionnaire-based study with a single assessment (no follow-up). Adults (≥18 years) with intracranial meningioma diagnosed on imaging and/or confirmed surgically will be invited. Exclusion criteria include inability to complete questionnaires independently, insufficient French comprehension, pregnancy/breastfeeding, legal deprivation of liberty, and individuals under compulsory psychiatric care.

Participants receive study information (in clinic when applicable, otherwise by email) and access a secure REDCap link. Non-opposition is recorded online prior to questionnaire completion. Participants complete MQOL-FR (70 items), EQ-5D-5L, and FACT-Br. The total completion time is estimated at 30-45 minutes; completion may be split into multiple sessions using a REDCap-provided access code. Data are collected directly in REDCap and stored in pseudonymized form.

Primary outcome is psychometric performance of MQOL-FR, including dimensionality/structural validity, internal consistency (e.g., Cronbach's alpha), construct and convergent validity against EQ-5D-5L and FACT-Br, completeness rates, and floor/ceiling effects. Secondary objectives are descriptive and exploratory: to summarize MQOL-FR, EQ-5D-5L, and FACT-Br scores in the overall cohort and compare subgroups (e.g., WHO grade, sporadic vs progestin-associated, symptomatic vs asymptomatic, skull base vs convexity, tumor size, single vs multiple lesions, and management strategy). Exploratory modeling (ANCOVA/regression) will be used to assess factors associated with MQOL-FR scores. The targeted analyzable sample is 100 complete MQOL-FR responses; based on prior completion rates, approximately 238 patients will be contacted to achieve this target. In accordance with the collaboration with the original MQOL developers, de-identified score data may be shared for scientific purposes.

ELIGIBILITY:
Inclusion Criteria :

* Inclusion Criteria:
* Age ≥ 18 years
* Diagnosis of intracranial meningioma on imaging and/or confirmed by surgery

Exclusion Criteria:

* Pregnant or breastfeeding
* Individuals deprived of liberty by judicial/administrative decision or under compulsory psychiatric care
* Insufficient French language proficiency/comprehension
* Unable to complete the questionnaires independently
* Unable to express non-opposition to participation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults with intracranial meningioma, recruited through three sources to maximize heterogeneity: (1) patients seen in consultation at GHU Paris-Sainte-Anne; (2) members of the AMAVEA patient association informed by email; and (3) patients proposed by partner teams after a call for participation within the French Society of Neurosurgery Neuro-Oncology Club and Skull Base Club, contacted by email and invited to complete online questionnaires via REDCap.
Sampling Method: Non-Probability Sample
Enrollment: 238 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-09-02 (Estimated); Study Completion 2026-09-02 (Estimated)

PRIMARY OUTCOMES:
Meningioma Quality of Life Questionnaire - French version (MQOL-FR) : psychometric performance (structural validity, internal consistency, construct/convergent validity, completeness, floor/ceiling effects) | Single assessment at enrollment (one questionnaire session; participants may complete within up to 1 month after invitation).
  The MQOL-FR is the French translation of the Meningioma Quality of Life questionnaire (MQOL), a self-administered, meningioma-specific health-related quality-of-life instrument (70 items across 9 domains). Total score range: 0 to 100; higher scores indicate a better outcome (better quality of life).